CLINICAL TRIAL: NCT04004728
Title: Aavaliação do Tratamento de Telangiectasias Dos Membros Inferiores Com Laser 1064mm
Brief Title: Laser Treatment Of Leg Telangiectasias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Nelson Wolosker, Principal Investigator, Associate Professor, MD, PhD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSR 0072/09
Record Dates: First submitted 2011-09-21; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Leg Veins
Keywords: laser; telangiectasias; leg veins; sclerotherapy
MeSH Terms: conditions — Telangiectasis

STUDY DESIGN:
Intervention Model Description: One leg laser ando the other sclerotherapy.
Masking Description: Blind photo evaluation.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- laser, leg veins, sclerotherapy (Other): to compare laser and sclerotherapy on treating leg veins
  Interventions: Procedure: 1064 Nd:YAG laser

INTERVENTIONS:
Procedure: 1064 Nd:YAG laser — 1064 laser - 135J 25ms spot 3mm GLicose - 75% - 3 ml

SUMMARY:
Is 1064 nm YAG Laser better than sclerotherapy to treat leg veins?

DETAILED DESCRIPTION:
Comparison between laser and sclerotherapy in the treatment of telangiectasias of legs.

ELIGIBILITY:
Inclusion Criteria:

* patients with leg telangiectasias

Exclusion Criteria:

* varicose veins
* DVT
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Changes analysis after treatments of leg telangiectasias´clearance through photography using a scale of improvement. | Analysis of photographic changes previous, and one week after treatment. Patient reanalysis after 1 and 3 months
  Patients are asked about the best method to treat leg veins after three treatments of laser and three treatments of sclerotherapy. Evaluation of the photographic improvement of the treated areas on a scale of 0 (no improvement) to 10 (complete cleaning of the vessels).
Changes analysis after treatments of leg telangiectasias´clearance using a questionnaire to classify the pain | 1 week after treatment
  Patients are asked about the best method to treat leg veins after three treatments of laser. All patients were asked to respond to a questionnaire classifying the pain (none, little, very painful or extremely painful).
Changes analysis after treatments of leg telangiectasias´clearance using a questionnaire to classify the cleaning of vessels | 1 week after treatment
  Patients are asked about the best method to treat leg veins after three treatments of laser. All patients were asked to respond to a questionnaire classifying the cleaning of vessels (poor, regular, good or excellent)
Changes analysis after treatments of leg telangiectasias´clearance using a questionnaire to classify the satisfaction with results | 1 week after treatment
  Patients are asked about the best method to treat leg veins after three treatments of laser. All patients were asked to respond to a questionnaire classifying satisfaction with results (nothing, little or much

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Wolosker, MD, PhD, Study Director — Hospital das Clinicas, University of Sao Paulo
Locations (1):
- Vascular Surgery HCFMUSP, São Paulo, Brazil